CLINICAL TRIAL: NCT06629142
Title: Comparing Optimized Models of Primary And Specialist Services for Palliative Care: Pilot Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Principal Investigator, Scott Halpern, John M. Eisenberg Professor of Medicine, Epidemiology, and Medical Ethics & Health Policy, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 100917710; PLACER-2022C3-30553 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Seriously Ill Hospitalized Patients
Keywords: Palliative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standardized Usual Care (Active Comparator): Active control group, where moderately high-risk patients (e.g., with a 1-year mortality risk between 60% and 94%) will receive usual care. A specialist PC consult is ordered by default for the highest-risk patients (i.e., 1-year mortality risk ≥ 95%), unless clinicians cancel the order.
  Interventions: Behavioral: Standardized Usual Care
- Trained Generalist Palliative Care (Experimental): Generalist clinicians trained in PC domains receive an EHR-based alert to document whether or not they have addressed PC domains for moderately high-risk patients ('accountable justification intervention'). A specialist PC consult is ordered by default for the highest-risk patients unless clinicians cancel the order.
  Interventions: Behavioral: Default Order; Behavioral: Accountable Justification
- Specialist Palliative Care (Experimental): A specialist PC consult is ordered by default for all patients with a ≥ 60% 1-year mortality risk ('default order intervention'), unless clinicians cancel the order.
  Interventions: Behavioral: Default Order

INTERVENTIONS:
Behavioral: Default Order — A specialist PC consult is automatically ordered for patients meeting a certain threshold of 1-year mortality risk (dependent on arm). An EHR-based Our Practice Advisory (OPA) alert on Open Chart informs clinicians when the default order will become active, and how to cancel an order within 24 hours if they elect to do so.
  Arms: Specialist Palliative Care; Trained Generalist Palliative Care
Behavioral: Accountable Justification — An EHR-based Our Practice Advisory alert asks generalist clinicians to self-report whether they have provided primary PC by clicking which of 4 key PC domains they have addressed or to provide a brief justification as to why not.
  Arms: Trained Generalist Palliative Care
Behavioral: Standardized Usual Care — Moderately high-risk patients (e.g., with a 1-year mortality risk between 60% and 94%) will receive usual care. For very high-risk patients (e.g., with a 1-year mortality risk of ≥ 95%), an EHR-based Our Practice Advisory (OPA) alert on Open Chart informs clinicians when the default order will become active, and how to cancel an order within 24 hours if they elect to do so.
  Arms: Standardized Usual Care

SUMMARY:
Palliative care (PC) seeks to reduce suffering and improve quality of life for patients with serious illnesses and their families. National guidelines recommend that clinicians either provide palliative care themselves (generalist PC) or consult experts (specialist PC) as a standard part of serious illness care. This feasibility pilot study will be conducted with 6 hospitals at two large U.S. health systems and enroll 540 seriously ill hospitalized patients. Eligibility is determined by a mortality prediction score where enrolled patients have at least a 60% risk of dying within 1 year. Enrollment assessment occurs as close as possible to 36 hours post admission. In this cluster-randomized trial, the 6 hospitals will be randomized to 3 arms: (1) standardized usual care, (2) trained generalist PC, or (3) specialist PC. Generalists are trained using the Center to Advance Palliative Care (CAPC) online trainings. The pilot study will only measure process outcomes to assess the feasibility of a larger clinical trial (e.g., are the interventions working as intended). This pilot feasibility study is the precursor to a much larger pragmatic, hybrid effectiveness-implementation parallel-cluster RCT that will assess the comparative effectiveness of triggering generalist PC and specialist PC on several patient-centered outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older; AND
* Predicted 1-year mortality risk of 60% or greater; AND
* Admitted to a study hospital.

Exclusion Criteria:

- Patients who die or have an active or completed discharge order prior to enrollment time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1208 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Appropriate Firings of All Our Practice Advisory (OPA) Interventions | 36 to 60 hours post admission
  Percentage of all Intervention Our Practice Advisory (OPAs) that fired in the correct time window for patients with mortality risk thresholds eligible for each intervention.

SECONDARY OUTCOMES:
Patient-Reported Outcome (PRO) Survey Response Rate at 1 month | Enrollment - 1 month post-discharge
  Percentage of 1-month PRO surveys completed by alive patients or their surrogate proxies
PRO Survey Response Rate at 3 months | Enrollment - 3 months post-discharge
  Percentage of 3-month PRO surveys completed by alive patients or their surrogate proxies
Default Specialist PC Consults | 36 hours to 170 hours post admission
  Percentage of default specialist PC orders that resulted in an inpatient PC consult before hospital discharge
Default Specialist PC Order Cancellation Rate | 36 hours to 60 hours post admission
  Percentage of default specialist PC orders in which a generalist clinician indicated they did not want the order to proceed.
Inappropriate Our Practice Advisory (OPA) Firings | 0 to 60 hours post admission
  Percentage of all patient encounters in whom at least one Our Practice Advisory (OPA) fired inappropriately. This includes an OPA firing outside the allowed time window on a patient who is eligible, the firing of the wrong OPA on a patient who is eligible (e.g., firing of the Generalist PC OPA for a patient in the Specialist PC arm), and the firing of any OPA on a patient who is ineligible (e.g., who has an inappropriate mortality risk score or active discharge order at the time enrollment eligibility is assessed).
Generalist PC Training Completion | Baseline
  Percentage of clinicians eligible for CAPC palliative care training in the Generalist PC arm who complete the 4 required training modules. Partial completion (1-3 required modules) and completion of optional CAPC modules will be secondarily reported.
Generalist PC Domain Completion | 36 hours to 60 hours post admission
  Percentage of clinicians in the Generalist PC arm who say they are addressing patients' PC needs during the current encounter, and of those, the percentage who document at least 1 of 4 PC Domains in the EHR Our Practice Advisory Alert

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Courtright, MD, MS, Principal Investigator — University of Pennsylvania; Scott Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Kaiser Permanente Southern California, Pasadena, California
  - Trinity Health, Livonia, Michigan